CLINICAL TRIAL: NCT06326073
Title: Evaluation of the GCF Periostin, IL-17A and IL-17E Levels of Smoking and Non-smoking Periodontitis Patients Received Periodontal Treatment: Short-term Follow-up Study
Brief Title: Interaction Between Smoking, GCF Periostin, IL17A, IL17E and Non-surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sule Ozdogan, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OMUKAEK2019/324
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis; Smoking
Keywords: non surgical periodontal therapy; smoking; periostin; IL-17; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Intervention Model Description: The study included systemic healthy smokers(SP)(n:11) and non-smokers(P)(n:11) with periodontitis, smokers (SH)(n:11) and non-smokers(H)(n:11) with periodontal healthy individuals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I: SP (Experimental): smokers with periodontitis
  Interventions: Procedure: Non Surgical Periodontal Treatment
- Group II: P (Experimental): non-smokers with periodontitis
  Interventions: Procedure: Non Surgical Periodontal Treatment
- Group III: SH (No Intervention): smokers with periodontal healthy individuals
- Group IV: H (No Intervention): non-smokers with periodontal healthy individuals

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment — Phase 1 periodontal (full mouth debridement) treatment was applied to groups with periodontitis in one session.
  Arms: Group I: SP; Group II: P

SUMMARY:
It was aimed to evaluate the changes in the levels of Periostin, IL-17A and IL-17E cytokines in the gingival crevicular fluid (GCF) of periodontitis patients which non-surgical (Phase I) periodontal treatment applied to and their interactions with smoking. The study included systemic healthy smokers(SP)(n:11) and non-smokers(P)(n:11) with periodontitis, smokers (SS)(n:11) and non-smokers(S)(n:11) with periodontal healthy individuals Phase I periodontal treatment was applied to the groups with periodontitis. Before treatment (day 0), clinical measurements evaluating periodontal status were recorded and GCF samples were collected. GCF samples were collected from the same tooth regions on the 15th and 30th days after treatment and clinical measurements were repeated. GCF Periostin, IL-17A and IL-17E levels were determined by ELISA method. All data were evaluated statistically.

DETAILED DESCRIPTION:
The SH and H groups' patients were instructed to visit for routine controls without receiving any periodontal treatment. However, after the GCF sampling, patients in the SP and P groups received Non-surgical periodontal treatment(NSPT) included detailed oral hygiene instruction and reinforcement in conjunction with scaling and root planning as a full mouth debridement protocol in a single session They were instructed to refrain from using any chemicals, including mouthwash, to remove plaque.

The periodontitis patients received a follow-up call on the 15th and 30th days following treatment. The GCF sampling procedure was first repeated on the teeth from which a previous GCF sample had been taken. Then, values for the clinical examination parameters (PI, GI, BOP, PD, and CAL) were once again measured and recorded. Daily plaque care efficacy or deficiency was checked and/or reinforced at every recall. All these procedures were performed by a single investigator.

ELIGIBILITY:
Inclusion Criteria:

* generalized stage 3 periodontitis or periodontally healthy;
* smoker ((≥10 cigarettes/day for >5 years) or nonsmoker (never smoked in their lifetime);
* not have received any periodontal treatment in the last 6 months, took any antibiotics, anti-inflammatory drugs regularly and for female subjects, not to be pregnant, lactating, or menopause.

Exclusion Criteria:

* Under 18 years of age
* Those with a systemic disease
* Cancer patients, those with a history of chemotherapy and radiotherapy
* Pregnant and breastfeeding women
* Those who smoke less than 10 cigarettes a day and those who quit smoking
* Having received orthodontic treatment in the last 6 months
* Using antibiotics, anti-inflammatory or any medication in the last 6 months
* Those who do not consent voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Periostin levels | 0-15-30 days
  The effect of non-surgical periodontal treatment in gingival crevicular fluid periostin levels
Evaluation of IL-17A levels | 0-15-30 days
  The effect of non-surgical periodontal treatment in gingival crevicular fluid IL-17A levels
Evaluation of IL-17E levels | 0-15-30 days
  The effect of non-surgical periodontal treatment in gingival crevicular fluid IL-17E levels

SECONDARY OUTCOMES:
Interaction Between Smoking and GCF Periostin, IL17A, IL17E levels | 0-15-30 days
  Comparisons between groups were made to evaluate the effect of smoking on non-surgical periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Muge Luftioglu, Study Director — Ondokuz Mayıs Universitesi
Locations (1):
- Ondokuz Mayıs University Faculty of Dentistry Department of Periodontology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT06326073/Prot_SAP_000.pdf